CLINICAL TRIAL: NCT07321405
Title: Non Invasive Hemodynamic Assessment of Cardiac Output and Stroke Volume in Septic Shock Patients
Brief Title: Assessment of Cardiac Output and Stroke Volume in Septic Shock Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Osman Mohamed Osman Khalaf, resident physician, Assiut University
Other Study IDs: COP and SV in septic shock
Record Dates: First submitted 2025-11-24; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- septic shock patients: echocardiography and electrical cardiometry will be applied to these patients
  Interventions: Device: echocardiogram; Device: Electrical cardiometry

INTERVENTIONS:
Device: echocardiogram — Transthoracic echocardiography (TTE) is the gold standard for non-invasive bedside assessment of CO and SV, providing precise evaluation of cardiac structure and flow. However, TTE requires operator expertise, can be time-consuming, and may be limited by patient-specific factors.
Device: Electrical cardiometry — Electrical cardiometry (EC) is an emerging non-invasive bio-impedance technique offering continuous monitoring with easier application and less operator dependency. Despite its advantages, EC's accuracy and reliability in critically ill septic patients require further validation.

SUMMARY:
The aim of this research is to compare the accuracy and reliability of electrical cardiometry versus transthoracic echocardiography in measuring cardiac output and stroke volume in patients with septic shock, to evaluate the potential of EC as a non-invasive alternative for hemodynamic monitoring.

DETAILED DESCRIPTION:
Sepsis is a life-threatening condition caused by a dysregulated immune response to infection, leading to organ dysfunction. It remains a leading global cause of morbidity and mortality, often progressing rapidly to septic shock and multi-organ failure if not promptly diagnosed and treated.

The complex pathophysiology involves systemic inflammation, endothelial damage, and impaired tissue perfusion, making early recognition and hemodynamic stabilization vital for survival. Accurate monitoring of cardiac function plays a key role in managing septic patients.

Cardiac output (CO) and stroke volume (SV) are key hemodynamic parameters guiding therapy in critically ill patients, particularly those with pneumonia and septic shock, who experience severe circulatory and respiratory dysfunction contributing to their high mortality.

Transthoracic echocardiography (TTE) is the gold standard for non-invasive bedside assessment of CO and SV, providing precise evaluation of cardiac structure and flow. However, TTE requires operator expertise, can be time-consuming, and may be limited by patient-specific factors.

Electrical cardiometry (EC) is an emerging non-invasive bio-impedance technique offering continuous monitoring with easier application and less operator dependency. Despite its advantages, EC's accuracy and reliability in critically ill septic patients require further validation.

Currently, hemodynamic monitoring mainly relies on clinical assessment combined with intermittent TTE, with invasive methods reserved for selective cases; EC holds potential as a simpler, safer alternative warranting further investigation.

ELIGIBILITY:
Inclusion Criteria: patients aged more than 18 years must be diagnosed with septic shock following the surviving sepsis campaign

-

Exclusion Criteria:

* patients aged less than 18 years pregnant women cases suffering cardiac diseases (heart failure, arrhythmia, moderate, and severe valvular disease) patients with poor quality echocardiographic images and measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients were aged more than 18 years diagnosed with septic shock following the surviving sepsis campaign
  -
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-10 (Estimated)

PRIMARY OUTCOMES:
to compare the accuracy and reliability of electrical cardiometry versus transthoracic echocardiography in measuring cardiac output in patients with septic shock. | 2026-2028
  to compare the accuracy and reliability of electrical cardiometry versus transthoracic echocardiography in measuring cardiac output in patients with septic shock.
cardiac output and stroke volume in septic shock patients | baseline
  comparison between accuracy and reliability in assessment of cardiac out put and stroke volume using echocardiogram vs electrical cardiometer
to compare the accuracy and reliability of electrical cardiometry versus transthoracic echocardiography in measuring stroke volume in patients with septic shock. | 2026-2028
  to compare the accuracy and reliability of electrical cardiometry versus transthoracic echocardiography in measuring stroke volume in patients with septic shock.

CONTACTS AND LOCATIONS:
Overall Officials: ahmed obeid allah, professor, Study Director — Assiut University; alaa abd elbadee, lecturer, Study Chair — Assiut University; mostafa hosney, lecturer, Study Chair — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Song W, Guo J, Cao D, Jiang J, Yang T, Ma X, Yuan H, Wu J, Guan X, Si X. Comparison of noninvasive electrical cardiometry and transpulmonary thermodilution for cardiac output measurement in critically ill patients: a prospective observational study. BMC Anesthesiol. 2025 Mar 13;25(1):123. doi: 10.1186/s12871-025-03005-1. PMID 40082773
- See also: https://pubmed.ncbi.nlm.nih.gov/40082773/ — https://pubmed.ncbi.nlm.nih.gov/40082773/